CLINICAL TRIAL: NCT07203937
Title: Effects of Combined Robotic and Conventional Lower Limb Rehabilitation on Quality of Life, Depression, Anxiety, and Fatigue After Stroke: A Randomized Controlled Trial
Brief Title: Effects of Robotic Rehabilitation on Quality of Life, Mood, and Fatigue After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Gunes Akinci (Other)
Responsible Party: Sponsor-Investigator, Meltem Gunes Akinci, Assistant Professor, Department of Physical Medicine and Rehabilitation, Pamukkale University Faculty of Medicine, Denizli, Türkiye, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-695640
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Post-stroke Depression; Post-stroke Anxiety; Post-stroke Fatigue; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional + Robotic Rehabilitation (Experimental): Participants in this arm will receive conventional rehabilitation (stretching, strengthening, balance and coordination, postural control, and gait training) 5 days per week for 6 weeks, combined with robotic-assisted gait training using the RoboGait® device 2 days per week for 6 weeks.
  Interventions: Device: RoboGait® Robotic Gait Training
- Conventional + Treadmill Training (Active Comparator): Participants in this arm will receive conventional rehabilitation (stretching, strengthening, balance and coordination, postural control, and gait training) 5 days per week for 6 weeks, combined with treadmill walking training 2 days per week for 6 weeks. The treadmill sessions will be matched in duration to the robotic gait training sessions of the experimental group.
  Interventions: Device: Treadmill Walking Training

INTERVENTIONS:
Device: RoboGait® Robotic Gait Training — RoboGait® is a robotic lower limb orthosis system with adjustable dynamic body weight support, synchronized treadmill, and biofeedback software. Participants will receive robotic-assisted gait training 2 days per week for 6 weeks, in addition to conventional rehabilitation 5 days per week.
  Other Names: Robotic-Assisted Rehabilitation; Robotic-Assisted Walking Exercise
  Arms: Conventional + Robotic Rehabilitation
Device: Treadmill Walking Training — Participants will receive treadmill walking sessions 2 days per week for 6 weeks, combined with conventional rehabilitation 5 days per week. The treadmill sessions will be matched in duration and intensity to the robotic training sessions in the experimental arm.
  Other Names: Treadmill-based gait training
  Arms: Conventional + Treadmill Training

SUMMARY:
Stroke is a major cause of long-term disability and is often associated with reduced quality of life, depression, anxiety, and fatigue. Rehabilitation plays a key role in recovery, and robotic-assisted gait training provides intensive, repetitive, and individualized therapy. However, its effects on psychological outcomes and quality of life are not fully established.

This randomized controlled trial will compare conventional rehabilitation combined with robotic-assisted gait training to conventional rehabilitation combined with treadmill training in stroke survivors. Both groups will receive treatment 5 days per week for 6 weeks.

Assessments will be conducted at baseline, after 6 weeks of treatment, and at 3 months after treatment. The primary outcome is quality of life. Secondary outcomes include depression, anxiety, and fatigue. The results of this study will provide new evidence on the benefits of robotic rehabilitation for improving both physical and psychological well-being after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* History of ischemic or hemorrhagic stroke at least 3 months prior to enrollment
* Mini Mental State Examination (MMSE) score of 24 or higher
* Modified Ashworth Scale score < 2 in the lower extremities

Exclusion Criteria:

* Severe cognitive or communication impairment
* Mobility limitations due to joint contracture or deformity
* Presence of open wounds or pressure ulcers
* Uncontrolled hypertension or orthostatic hypotension
* Severe cardiovascular disease, heart failure, cancer, or significant pulmonary disease
* High fracture risk due to severe osteoporosis
* Ambulation difficulty caused by lower extremity musculoskeletal disorders
* Severe psychosis or neurosis
* Modified Ashworth Scale score > 3 in the lower extremities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Stroke-Specific Quality of Life Scale (SS-QoL) | Baseline (T0), 6 weeks post-treatment (T1), and 3 months post-treatment (T2)
  The Stroke-Specific Quality of Life Scale (SS-QoL) is a validated 49-item patient-reported questionnaire assessing 12 domains including mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality. Higher scores indicate better quality of life. The primary endpoint is the change in SS-QoL score from baseline to 3 months after treatment.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline (T0), 6 weeks post-treatment (T1), and 3 months post-treatment (T2)
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire evaluating fatigue severity. Each item is scored from 0 to 7, with higher mean scores indicating greater fatigue.
Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale | Baseline (T0), 6 weeks post-treatment (T1), and 3 months post-treatment (T2)
  The HADS-Anxiety subscale consists of 7 items rated on a 4-point Likert scale. Scores range from 0-21, with higher scores indicating greater anxiety.
Hospital Anxiety and Depression Scale (HADS) - Depression Subscale | Baseline (T0), 6 weeks post-treatment (T1), and 3 months post-treatment (T2)
  The HADS-Depression subscale consists of 7 items rated on a 4-point Likert scale. Scores range from 0-21, with higher scores indicating greater depressive symptoms.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and institutional data protection policies. Only summary results will be disseminated through scientific publications and conference presentations.

REFERENCES:
- [Background] Haolin T, Yuanbin Y, Hu Z, Wenjing Z, Jing Z, Jingfeng T, Long HE, Xuechao LI, Qinxuan S, Mei S. Efficacy of Daoyin combined with lower limb robot as a comprehensive rehabilitation intervention for stroke patients: a randomized controlled trial. J Tradit Chin Med. 2024 Jun;44(3):530-536. doi: 10.19852/j.cnki.jtcm.20240322.002. PMID 38767637
- [Background] den Brave M, Beaudart C, de Noordhout BM, Gillot V, Kaux JF. Effect of robot-assisted gait training on quality of life and depression in neurological impairment: A systematic review and meta-analysis. Clin Rehabil. 2023 Jul;37(7):876-890. doi: 10.1177/02692155231152567. Epub 2023 Jan 22. PMID 36683416
- [Background] Mustafaoglu R, Erhan B, Yeldan I, Gunduz B, Tarakci E. Does robot-assisted gait training improve mobility, activities of daily living and quality of life in stroke? A single-blinded, randomized controlled trial. Acta Neurol Belg. 2020 Apr;120(2):335-344. doi: 10.1007/s13760-020-01276-8. Epub 2020 Jan 28. PMID 31989505